CLINICAL TRIAL: NCT04233021
Title: A Phase II, Multi-centre Study, to Evaluate the Efficacy and Safety of Osimertinib Treatment for Patients with EGFR-mutated Non-small Cell Lung Cancer (NSCLC) with Brain or Leptomeningeal Metastases
Brief Title: Study of Osimertinib in Patients with a Lung Cancer with Brain or Leptomeningeal Metastases with EGFR Mutation
Acronym: ORBITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1804
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Leptomeningeal Metastasis; Brain Metastases; EGFR Activating Mutation
Keywords: IFCT; NSCLC; EGFR
MeSH Terms: conditions — Meningeal Carcinomatosis; Brain Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib (Experimental): Osimertinib 80 mg/d
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 80 mg/d

SUMMARY:
Treatment of non-small cell lung cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) mutation is mainly based on tyrosine kinase inhibitors (TKIs) targeting EGFR. 1st or 2nd generation inhibitors have been shown to be superior to chemotherapy in terms of Progression-Free Survival (PFS) when used as 1st line treatment.

In case of progression at several metastatic sites, systemic treatment will be considered and will depend on the presence of the TKI resistance mutation, the T790M mutation. In the presence of the T790M mutation, osimertinib is superior to chemotherapy in terms of progression-free survival, while in the absence of the T790M mutation, platinum salt chemotherapy is recommended. In case of local progression, treatment of the site in progression by radiotherapy and/or surgery is considered. As these local treatments can cause long-term adverse effects, systemic treatments are increasingly being considered in this indication.

Brain and leptomeningeal metastases are the most frequent isolated site of progression in EGFR mutated patients treated with TKI. The high frequency of isolated cerebral and leptomeningeal progression is a consequence of the lower diffusion of 1st and 2nd generation TKIs in the central nervous system (CNS). Osimertinib is a 3rd generation TKI that has the particularity of overcoming the T790M mutation and having greater brain penetration than 1st or 2nd generation TKIs, which could make it an attractive therapeutic option in the event of brain progression or leptomeningeal progression. However, its efficacy in patients with cerebral or leptomeningeal metastases is still poorly understood.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with NSCLC (histological or cytological diagnosis) stage IV (8th UICC TNM edition, 2017).
2. Patients with brain and/or leptomeningeal metastases. For cohort 1, the diagnosis of leptomeningeal metastasis requires either 1) detection of cancer cell or EGFR mutation in the CSF, or 2) presence of both clinical and neuro-imaging findings typical of LM, according to EANO-ESMO criteria.
3. Presence of an activating EGFR mutation. The following mutations are considered to be activating: L858R, exon 19 deletions, exon 19 insertions, L861Q, G719X. The inclusion of patients with other mutations should be discussed on a case-by-case basis with IFCT.

   The presence of co-mutations on an oncogenic driver should be discussed with the IFCT before inclusion of the patient.
4. Testing for T790M mutation in circulating tumour DNA or tumour tissue sample at progression on the last treatment received before inclusion.
5. Maximum lines of anti-cancer treatment received before inclusion:

   * For Cohort 1, patients could have been previously treated with maximum 3 lines of anti-cancer treatment.
   * For cohort 2, patients could have been previously treated with maximum 1 line of anti-cancer treatment.

   In case of previous chemotherapy, a wash-out period of 28 days will be applied. If there was any prior therapy with an investigational agent, a washout period of five half-lives of the compound or 3 months, whichever is greater, is needed.
6. Patient having recovered from all grade ≤ 1 toxicities related to previous anticancer therapies (CTCAE v 5.0) except for alopecia, platinum-therapy-related neuropathy (where ≤2 is allowed).

8. Presence of at least one evaluable lesion not previously irradiated according to RECIST 1.1. For cohort 2, presence of one CNS evaluable lesion not previously irradiated according to RECIST 1.1.The radiological assessment has to be done within the timelines indicated.

9. Age of at least 18 years old. 10. Performance status (PS) 0 to 2 (ECOG) except for patients with leptomeningeal carcinomatosis (cohort 1) a PS 3 is authorised.

11. Patient with a life expectancy of ≥ 6 weeks for cohort 1 and ≥ 12 weeks for cohort 2.

12. Haematological function:

* Absolute number of neutrophils ≥ 1.5 x 109/L;
* Platelets ≥ 100 x 109/L;
* Haemoglobin ≥ 9 g/dL (transfusions to maintain or exceed this value are accepted).

  13. Hepatic function:
* Total bilirubin ≤ 1.5 x UNL (Upper Normal Limit) or ≤ 3 x UNL in case of documented Gilbert's syndrome or liver metastases;
* AST / ALT < 2.5 x UNL if no liver metastases or < 5 x UNL in case of liver metastases.

  14. Renal function: Creatinine ≤1.5 x UNL. If creatinine > 1.5 x UNL, Creatinine clearance must be ≥ 50 mL/min (Cockroft or MDRD or CKD-epi) 15. Coagulation:
* International Normalized Ratio (INR) ≤ 1.5 ;
* Prothrombin Ratio (PR) ≤ 1.5 x UNL. 16. Patient having signed an informed consent form prior to any study specific procedure 17. Patient able, according to the investigator, to comply with study requirements, 18. Patient covered by a national health insurance 19. Female subjects should be using highly effective contraceptive measures during the study and 2 months after discontinuing osimertinib (highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly), and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation 20. Male subjects should be willing to use highly effective barrier contraception during the study and for 4 months after discontinuing osimertinib

Exclusion Criteria:

1. Small cell lung cancer histology (SCLC) or tumours with mixt histology including a SCLC component.
2. Previous treatment with osimertinib or another 3rd generation EGFR inhibitor.
3. Previous treatment with any EGFR TKI (cohort 2 only)
4. Brain progression requiring whole brain radiation without delay.
5. Local treatments (neurosurgical or stereotactic treatment) for brain metastases performed less than 2 weeks prior to enrolment.
6. Local brain treatment scheduled during study treatment.
7. Patient who received radiotherapy including the lung fields ≤ 4 weeks before enrolment or patient who has not recovered from radiotherapy-induced toxicities. For all other body sites (including radiotherapy on thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks before enrolment or who have not recovered from radiotherapy-induced toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks before enrolment is authorised.
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec using the screening clinic ECG machine derived QTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block and second degree heart block).
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
9. Active malignant disease other than NSCLC.
10. Previous or active cancer within the previous 3 years (except for treated carcinoma in situ of the cervix or basal cell skin cancer).
11. Others on-going anti-cancer treatment (including hormone therapy).
12. Major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic) during the 4 weeks before enrolment or patient who has not recovered from the side effects of such as procedure.
13. Current severe infectious disease or fever > 38.5°C or evidence of any other pathology, degradation of organic or neurological functions, result of the physical examination or laboratory tests leading to suspect disease or a condition contra-indicating the use of the study treatment, which can impair the patient's compliance to the protocol conditions or expose to any possible risk of complications related to treatment.
14. Clinically significant heart disease (e.g. active): stroke or myocardial infarction in the 6 months prior to inclusion, unstable angina, congestive heart failure grade > II according to New York Heart Association (NYHA) parameters, or cardiac arrhythmia requiring specific treatment during the study which could interfere with study compliance or which is not controlled by a treatment.
15. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).Active infection will include any patients receiving treatment for infection. Participants with a resolved or chronic infection HBV are eligible if they are:

    * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG] or
    * Positive for HBsAg, negative for HBeAg but for > 6 months have had transaminases levels below ULN and HBV DNA levels below 2000 IU/mL (i.e., are in an inactive carrier state).
16. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
17. History of hypersensitivity to any of the active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
18. Currently receiving (or unable to stop use at least 3 week prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (see Appendix 2). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
19. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
20. Patient who is subject to legal protection or who is unable to express his will.
21. Patient with a deficiency preventing complete understanding of the study requirements.
22. Patient having already been included and treated in this study or in another clinical trial (except for biological trials consisting of taking samples only).
23. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  Objective Response Rate at 6 months using EANO-ESMO criteria (cohort 1) and RECIST1.1 criteria (cohorts 2)

SECONDARY OUTCOMES:
Overall Survival | About 24 months
  Time from enrollment until death due to any cause
Progression-free survival | About 24 months
  Time from enrollment to first observation of progression (EANO-ESMO criteria (cohort 1) and RECIST1.1 criteria (cohorts 2) or date of death (from any cause)
CNS Progression-free survival | About 24 months
  Time between the date of randomization and the first date of documented CNS progression, or death in the absence of progression due to any cause, whichever occurs first.
Incidence, type and severity of adverse event | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (about 24 months)
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Evaluate the Quality of life | From time of randomisation through treatment period (about 24 months)
  EORTC QLQ-C30-LC13 (Qualify of Life Questionnaire C30 and Lung Cancer 13) questionnaire
Evaluate the Quality of life | From time of randomisation through treatment period (about 24 months)
  QLQ BN20 (Brain Neoplasm N20) questionnaire
CNS Overall response Rate (ORR) | 6 months
  the percentage of subjects who have a best overall CNS response of Complete CNS Response (CR) or Partial CNS Response (PR) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: David PLANCHARD, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique; Franck MORIN, Study Director — Intergroupe Francophone de Cancerologie Thoracique
Locations (36):
- France (36):
  - Centre Hospitalier Aix-Pertuis, Aix-en-Provence
  - CHU Amiens - Groupe Hospitalier Sud, Amiens
  - Centre Paul Papin, Angers
  - Hôpital privé d'Antony, Antony
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Besançon - Hôpital J. MINJOZ, Besançon
  - Groupe Hospitalier Saint André, Bordeaux
  - AP-HP Hôpital Ambroise Paré, Boulogne
  - CHU Côte de Nacre, Caen
  - Hôpital Louis Pasteur, Colmar
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Hôpital du Bocage, Dijon
  - Chu Grenoble, Grenoble
  - Centre Hospitalier Général, Le Mans
  - Hôpital Calmette, Lille
  - CHU Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - Marseille Hôpital Nord, Marseille
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Régional - Hôpital de la Source, Orléans
  - AP-HP Hôpital Cochin, Paris
  - AP-HP Hôpital Bichat, Paris
  - Centre Hospitalier Général - Pau, Pau
  - Lyon - URCOT Centre Hospitalier Universitaire, Pierre-Bénite
  - CHU de la Réunion - Site Felix Guyon, Saint-Denis
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - CHU de La Réunion-Site Sud, Saint-Pierre
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - HIA Sainte-Anne, Toulon
  - Hôpital Larrey, Toulouse
  - CHU Bretonneau, Tours
  - Valenciennes Clinique PRIV, Valenciennes
  - Centre Hospitalier de Villefranche-sur-Saône, Villefranche-sur-Saône
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: IFCT Website — https://www.ifct.fr/index.php/fr/la-recherche/item/2169-ifct-1804-orbital